CLINICAL TRIAL: NCT06454071
Title: Relationship Between Immunologic Changes and Recovery-related Factors in the Recovery Process of Elderly Colon Cancer Patients
Brief Title: Immunologic Changes and Recovery-related Factors in Elderly Colon Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Soonchunhyang UH
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Cancer of Colon; Interleukins; Aged
MeSH Terms: conditions — Colonic Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: The entire number of patients was divided into elderly and non-elderly groups based on the age of 70. 29 patients were assigned in elderly group, and 46 patients were assigned in non-elderly group. Preoperative blood sampling including WBC, lymphocyte, neutrophil, albumin, globulin was performed for all patients. In case of participants, investigators added the additional blood tests including immunologic markers including Interleukin-6 and Natural killer cell. These blood tests including immunologic markers were conducted before surgery, on the third day following surgery, and on the first outpatient visit day (approximately 21 days after surgery)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interleukin6 (Other): Immunologic tests including Interleukin 6 were conducted before surgery, on the third day following surgery, and on the first outpatient visit day (approximately 21 days after surgery). The IL-6 tests were carried out in our hospital.
  Interventions: Other: Blood test
- NK cell (Other): Immunologic tests including Nk cell were conducted before surgery, on the third day following surgery, and on the first outpatient visit day (approximately 21 days after surgery). The NK cell tests were carried out in our hospital. Peripheral blood mononuclear cells were evaluated using flow cytometry via fluorochrome-conjugated antibodies against a number of NK cell receptors.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Immunologic tests including Interleukin 6 were conducted before surgery, on the third day following surgery, and on the first outpatient visit day (approximately 21 days after surgery). The IL-6 tests and NK cells were carried out in our hospital.

SUMMARY:
Colorectal cancer is one of the most frequent malignancies, with a rising proportion of elderly patients in an aging society. In this study, the investigators attempted to find out the relationship between immunologic factors and recovery using various parameters impacting the treatment in elderly patients.

DETAILED DESCRIPTION:
In prospective study, total 75 patients who received radical resection for colon cancer between September 2023 and February 2024 at Asan Medical Center was involved. Investigators included colon cancer patients treated with surgery, diagnosed with adenocarcinoma histologically and having information regarding preoperative status with abdominopelvic CT. Routine blood sampling and Immunologic tests including interleukin-6 (IL-6) and natural killer cell (NK cell) were performed at preoperative day, post operative 3rd day (POD#3), and outpatient clinic day (about postoperative 21th day (POD#21)). Investigators attempted to assess the patients' subjective health level using a simple questionnaire, EuroQol group- 5 dimension- 3 level (EQ-5D-3L). The sarcopenia was evaluated by the artificial intelligence software system and defined as an SMI < 41cm2/m2 in women and SMI < 43 cm2/m2 in men with a body mass index (BMI) < 25kg/m2, and < 53 cm2/m2 in men with a BMI ≥ 25 kg/m2.

In this study, primary end point was recovery represented by hospital stay defined as the day from operation to discharge and readmission within 30days after discharge. Secondary end point was EQ-5D-3L (only in prospective cohort). 'Recovery' was evaluated by hospital stay and readmission within 30 days after discharge. Analyses of clinicopathological characteristics of categorical variables and continuous variables were conducted using the chi-square test and t-test, respectively. A multivariable analysis with Cox proportional hazards model was used to compare risk factors associated with postoperative hospital day including NLR, AGR, albumin, BMI and sarcopenia. Investigators conducted an analysis including variables that have been proven to be related to the immune system or recovery in previous studies or that are suspected to be clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* colon cancer patients treated with surgery
* diagnosed with adenocarcinoma histologically
* having information regarding preoperative status with abdominopelvic CT

Exclusion Criteria:

* familial colorectal cancer
* malignancies other than adenocarcinoma
* inflammatory bowel disease-associated cancer
* recurrence
* metastasis

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Differences of recovery in between elderly and elderly patients | up to 1 month
  The primary end point was' recovery' represented by hospital stay. Investigators evaluated 'Recovery' by hospital stay and readmission within 30 days after discharge. Investigators categorized the patients who had a shorter-than-average hospital stay as 'fast' group, and patietns who had a longer-than-average hospital stay or readmitted within 30 days after discharge rated their recovery as 'slow' group.

CONTACTS AND LOCATIONS:
Overall Officials: Byeo Lee Lim, Dr, Study Director — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided